CLINICAL TRIAL: NCT00666861
Title: Understanding the Acute Effects of Prolonged Sedentary Behaviour (Sitting) on Post-meal Glucose and Lipids - A Pilot Study
Brief Title: Type 2 Diabetes and Exercise - A Pilot Study
Status: Terminated | Type: Observational
Why Stopped: Pilot study superseded by a larger NHMRC funded trial
Sponsor: Bayside Health (Other Government)
Collaborators: International Diabetes Institute, Australia (Other); Baker Heart Research Institute (Other)
Responsible Party: Assoc/Prof Bronwyn Kingwell - Executive Director Science Policy and Head, Clinical Physiology, Baker Heart Research Institute
Other Study IDs: 290/07
Record Dates: First submitted 2008-04-23; First posted 2008-04-25 (Estimated); Last update posted 2009-07-30 (Estimated); Status verified 2009-07

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma samples
Oversight: Data Monitoring Committee: No

SUMMARY:
A randomised, cross-over trial targeting a small sample of older (age 45-65 years) overweight adults with type 2 diabetes the aims of this pilot study are to:

1. Determine the feasibility of investigating the acute effects of prolonged sedentary behaviour (sitting) in this target group.
2. Compare the acute effects of a single prolonged (8 hour) bout of sedentary behaviour (sitting) on glucose and triglyceride concentrations and key muscle and adipose regulatory enzymes to a similar bout of sedentary behaviour combined with intermittent bouts of light-intensity activity.

DETAILED DESCRIPTION:
The proposed study will involve a randomised cross-over experimental trial conducted in the laboratory setting in older overweight adults with type 2 diabetes. Participants will receive both of the acute testing conditions in a randomised manner.

Study design: Randomised cross-over pilot trial of 20 overweight/obese older adults with diet-controlled type 2 diabetes involving 2 acute treatment conditions, with a one-week wash-out period between testing conditions (Figure 1 a).

Setting: Acute, supervised laboratory setting within the Alfred and Baker Heart Institute Medical Unit.

Outcomes: We will measure acute responses in laboratory-measured plasma glucose & triglyceride levels (every 60 mins) and glucose concentrations determined from continuous glucose monitoring (CGMS).

ELIGIBILITY:
Inclusion Criteria:

1. Diet controlled Diabetes
2. Overweight (BMI > 27 kg/m2 but <50 kg/m2)

Exclusion Criteria:

1. Hypoglycaemic Agents
2. Lipid Lowering Agents

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Type 2 Diabetes
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2008-04; Primary Completion 2008-10 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bronwyn A Kingwell, PhD, Principal Investigator — Baker Heart Research Institute
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia